CLINICAL TRIAL: NCT03987334
Title: Effects of Virtual Reality Motor Control Rehabilitation in Neck Pain Subjects
Brief Title: Virtual Reality Rehabilitation in Neck Pain Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Sandro Iannaccone, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR-NECKPAIN
Record Dates: First submitted 2019-05-23; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Neck Pain; Chronic Pain; Whiplash
Keywords: Virtual Reality; Motor Control; Augmented Feedback; Chronic Neck Pain; Whiplash
MeSH Terms: conditions — Neck Pain; Chronic Pain; Whiplash Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (VRT) (Experimental): Subjects in the experimental group (VRT) will undergo 30 minutes of motor control exercises using a virtual reality-based sensorimotor rehabilitation provided using the Virtual Reality Rehabilitation System (VRRS) of Khymeia Group. The equipment includes a computer workstation connected to a 6 degrees of freedom (DOF) motion-tracking system (Polhemus G4, Vermont, US), a high-resolution LCD displaying the virtual scenarios on a large screen and a software processing the motion data coming: from the receiver of the sensors end-effectors placed on the sternum and on the head through a helmet. The system has been found to reliably record head position and cervical range of motion among asymptomatic people as well as persistent neck pain patients. The VRRS allows the participant to perform the requested motor tasks, while the movement of the system's end-effector is simultaneously represented in a virtual scenario.
  Interventions: Other: Virtual Reality Treatment
- Control Group (CT) (Active Comparator): Control group (CT) subjects will undergo the same treatment of VRT subjects in terms of intensity, time and type, but with the VR turned off.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Virtual Reality Treatment — Experimental Group (VRT) subjects will undergo Virtual Reality Motor Control exercises based on augmented feedback of their performance.
  Other Names: Virtual Reality Motor Control Rehabilitation; Virtual Reality Augmented Feedback; Virtual Reality Rehabilitation System
  Arms: Experimental Group (VRT)
Other: Control Group — Control Group (CT) subjects will undergo the same treatment of VRT subjects in terms of intensity, time and type, but with the VR turned off.
  Other Names: Motor Control Rehabilitation
  Arms: Control Group (CT)

SUMMARY:
VR-NECKPAIN is a two-arm, monocentric, single-blind, randomized controlled trial in Neck Pain patients.

The entire treatment consist in 12 sessions, each during 45 minutes, twice a week for 6 consecutive weeks.

Subjects will be evaluated ad baseline (T0) and after six weeks of rehabilitation (T1). There will also be a 3 months Follow-Up assessment (T2).

The total duration of study participation for each subject will be approximately 19 weeks, including evaluation at T0, treatment and evaluation at T1 and T2.

Individuals in the experimental group (VRT) will undergo a virtual reality-based sensorimotor rehabilitation. Control group (CT) subjects will undergo the same rehabilitation of VR subjects, in terms of intensity, time and type, but with the virtual reality turned off.

DETAILED DESCRIPTION:
VR-NECKPAIN is a monocentric, single-blind, randomized controlled trial in Neck Pain patients.

Subjects will receive rehabilitation treatment twice a week, for six consecutive weeks. Subjects will be evaluated ad baseline (T0) and after six weeks of rehabilitation (T1). Also there will be a 3 months Follow-Up assessment (T2).

The total duration of study participation for each subject will be approximately 19 weeks, including evaluation at T0, treatment and evaluation at T1 and T2.

Individuals in the experimental group (VRT) will undergo a virtual reality-based sensorimotor rehabilitation. Control group (CT) subjects will undergo the same rehabilitation of VR subjects, in terms of intensity, time and type, but with the virtual reality turned off.

The study is conducted from March 2019 and the conclusion is planned to March 2023.

Patients with Neck Pain will be enrolled at the Department of Rehabilitation and Functional Recovery of San Raffaele Hospital, via Olgettina 60, Milan.

The treatment will last 45 minutes, 2 sessions per week for a total of 6 weeks. The first 15 minutes of treatment will consist, for each group, in manual therapy treatment, such as mobilization, manipulation, trigger-points treatment, tailored on the individual.

Subjects in the experimental Group (VRT) will undergo 30 minutes of motor control exercises using a virtual reality-based sensorimotor rehabilitation provided using the Virtual Reality Rehabilitation System (VRRS) of Khymeia Group. The equipment includes a computer workstation connected to a 6 degrees of freedom (DOF) motion-tracking system (Polhemus G4, Vermont, US), a high-resolution LCD displaying the virtual scenarios on a large screen and a software processing the motion data coming: from the receiver of the sensors end-effectors placed on the sternum and on the head through a helmet. The system has been found to reliably record head position and cervical range of motion among asymptomatic people as well as persistent neck pain patients.The VRRS allows the participant to perform the requested motor tasks, while the movement of the system's end-effector is simultaneously represented in a virtual scenario.

Control Group (CT) subjects will undergo the same treatment of VRT subjects in terms of intensity, time and type, but with the VR turned off.

In addition, all subjects will be educated in emphasizing self-management and return to normal function.

A blind assessor will be present in our study. In order to maintain him/her blind, treatments on patients will never take place in presence of the assessor.

Forty healthy subjects, matched for age and sex to the studied population, will also be enrolled in order to obtain normative data to compare with neck pain subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (18-70 years old);
* Neck Pain (Chronic Neck Pain or Whiplash);
* Normal vision or corrected vision.

Exclusion Criteria:

* Informed Consent negation;
* System infection or metabolic/neurological/muscular degenerative disorder;
* Cervical spinal pathology, fracture or surgery;
* Radiculopathy;
* Vestibular impairments;
* Epilepsy;
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The NDI is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. The NDI consists of 10 questions in various domains: Pain Intensity, Personal care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping and Recreation. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). Total score is reported on a 0-50 scale.

SECONDARY OUTCOMES:
Change in Numeric Rating Scale (NRS) | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The Numeric Rating Scale is a segmented numeric horizontal bar on which patients select a whole number (from 0 "no pain" to 10 "worst possible pain") that best reflects the intensity of their pain at rest and on movement. It has become a widely used instrument for pain screening and is ubiquitous as a screener in many health care environments.
Change in Neck and Pain Disability Scale (NPAD) | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The Neck and Pain Disability Scale is made by a 20 items measuring the intensity of pain and its interference with vocational, recreational, social and functional aspects of living and the presence and extent of associated emotional factors. Patients respond to each item by marking along a 10-cm visual analog scale. Item scores range from 0 to 5.
Change in Tampa Scale of Kinesiophobia (TSK) | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The Tampa Scale of Kinesiophobia is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The original questionnaire was developed to "discriminate between non-excessive fear and phobia among patients with chronic musculoskeletal pain". The scale was then found to be valid and reliable. Initially it was used in order to assess fear of movement related to chronic low back pain, but then it has been used for pain related to different parts of the body, including the cervical spine. The TSK is a self-completed questionnaire and the range of scores are from 17 to 68, where the higher scores indicate an increasing kinesiophobia.
Change in Active Range of Motion | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The distance and direction to which a bone joint can be extended. Range of motion is a function of the condition of the joints, muscles, and connective tissues involved.
Change in Conjunct Motion | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  Conjunct motion consists in cervical movements in the associated planes relative to the primary movement plane. It may reflect protective postural control strategies.
Change in Jerk Movements | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  Jerk Movements are the rate of changes in acceleration, a way to quantitatively evaluate smoothness of movements.
Changes in Joint Position Error (JPE) | Baseline (at recruitment/before intervention), Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The JPE will be recorded as the difference in head orientation between the start position (positioned vertically by a physiotherapist) and the position after a target catching in a 8 different circle-direction with movements of 20°.
Patient Global Impression of Change (P-GIC) | Post-Intervention (after 6 weeks rehabilitation), Follow-Up (after 3 months from completion of intervention)
  The Patient Global Impression of Change scale is recommended for use in chronic pain clinical trials as a core outcome measure of global improvement with treatment. The scale measures the change in patient's overall status since the beginning of the study on a scale of: 1 (very much improved); 2 (much improved); 3 (minimally improved); 4 (no change); 5 (minimally worse); 6 (much worse); and 7 (very much worse). This measure is a single-item rating by participants of their improvement with treatment during a clinical trial on a 7-point scale that ranges from 'very much improved' to 'very much worse' with 'no change' as the mid-point. The data provide a responsive and readily interpretable measure of participants' assessments of the clinical importance of their improvement or worsening over the course of a clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Ospedale San Raffaele, Milan, MI, Italy